CLINICAL TRIAL: NCT00234806
Title: Health-e-Access: A Study of Telemedicine in Primary Pediatric Care in Rochester, NY
Brief Title: Health-e-Access Telemedicine in Primary Pediatric Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: United States Department of Commerce (U.S. Federal Agency); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Kenneth McConnochie, Professor, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8858; AHRQ- R01 HS015165-02; MCHB- 1 R40MC03605-01-00
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Common Childhood Illnesses; Non-emergent Care
Keywords: telehealth; telemedicine

ARMS (2):
- Telemedicine intervention group (Experimental)
  Interventions: Other: Health-e-Access
- Control group (Placebo Comparator)
  Interventions: Other: Health-e-Access

INTERVENTIONS:
Other: Health-e-Access — telemedicine intervention

SUMMARY:
This study aims to take the existing model from the pilot of Telemedicine in Daycare and expand it to other suburban childcare centers and both urban and suburban elementary schools.

An assessment of the value of telehealth in the child programs will then be initiated to detail the impact of utilization and costs.

An assessment of the value of integrating telehealth into primary care practice will also be evaluated. The impact of continuity of care, well child visit rates, and immunization status will be among the various measures used in this evaluation.

DETAILED DESCRIPTION:
This involves estimating the impact of reduced absence due to illness on parents and their employers and estimating the value of a telehealth visit to these stakeholders. An interview instrument was developed to administer before experience with telehealth and again after a family has had experience with the program. In addition program attendance (childcare or school) records will be collected to document changes in absenteeism pre and post telehealth service implementation.

This study involves a before and after research design including both historical and concurrent controls comparing a detailed utilization of health services including telehealth visits, emergency department services and illness related office visits. Analyses will include center-level analyses of service utilization on a weekly basis pre and post as well as a child-level analyses including utilization before enrollment in a participating childcare center or school through program participation and, eventually, telehealth participation.

This is a descriptive observational study of the feasibility and acceptability of integrating telehealth service into 10 primary care pediatric practices. This study will document the integration process by maintaining a log of key communications relating to decision making (meeting minutes, memos, written agreements, protocols) and by interviewing key staff such as residents, nurse practitioners, attending physicians, staff nurses, and administrative leaders following the study period.

ELIGIBILITY:
Inclusion Criteria:

* All children at participating childcare centers and elementary schools.

Exclusion Criteria:

* Foster care children, children whose parents have refused participation, or children whose parents are unable to appropriately comprehend the program for any reason.

Ages: 6 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Actual)
Dates: Start 2000-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the impact of telehealth on utilization and cost of health care

SECONDARY OUTCOMES:
Evaluation of the feasibility and acceptability of integrating telehealth services into 10 primary care practices

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth McConnochie, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] McConnochie KM, Wood NE, Kitzman HJ, Herendeen NE, Roy J, Roghmann KJ. Telemedicine reduces absence resulting from illness in urban child care: evaluation of an innovation. Pediatrics. 2005 May;115(5):1273-82. doi: 10.1542/peds.2004-0335. PMID 15867035